CLINICAL TRIAL: NCT07345234
Title: Comparison Between Supine Mini Percutaneous Nephrolithotomy (PCNL) and Flexible Ureteroscopy (FURS) in Management of Lower Calyceal Stones 1-2 Centimeters With More Than 1000 Hounsfield Unit in School-Age Pediatric Patients
Brief Title: Comparison Between Supine Mini-PCNL and Flexible Ureteroscopy (FURS) for Dense Lower Calyceal Stones (1-2 cm) in School-Age Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shereef almegabar, Resident of Urology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU_MS814_2025
Record Dates: First submitted 2025-12-16; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Nephrolithiasis; Kidney Calculi; Urolithiasis
Keywords: pediatric; children; school-age; lower calyx; lower pole; renal stone; kidney stone; flexible ureteroscopy; high-density stone; mini percutaneous nephrolithotomy; laser lithotripsy
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi; Urolithiasis

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups to undergo either supine mini percutaneous nephrolithotomy with laser lithotripsy or flexible ureteroscopy with laser lithotripsy for management of dense lower calyceal renal stones.
Masking Description: This was an open-label study; participants and treating clinicians were aware of the assigned procedure. Outcome assessment was based on postoperative imaging and clinical follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine Mini Percutaneous Nephrolithotomy (Active Comparator): Participants underwent supine mini percutaneous nephrolithotomy for lower calyceal renal stones. A ureteral catheter was placed cystoscopically, renal access was obtained under fluoroscopic guidance with an 18-gauge needle, a guidewire was inserted, and tract dilation was performed up to 16 French followed by placement of a renal access sheath. Stones were fragmented using laser lithotripsy via a mini nephroscope. A double-J ureteral stent was placed, and a nephrostomy tube was left in place per protocol.
  Interventions: Procedure: Supine Mini Percutaneous Nephrolithotomy
- Flexible Ureteroscopy (Active Comparator): Participants underwent flexible ureteroscopy in the dorsal lithotomy position. After cystoscopy, a guidewire was advanced into the renal pelvis under fluoroscopic guidance. A digital flexible ureteroscope was used to access the kidney and visualize the stone. Stone fragmentation was performed using laser lithotripsy (dusting technique per protocol). A double-J ureteral stent was placed and scheduled for removal approximately 3 to 4 weeks after the procedure.
  Interventions: Procedure: Flexible Ureteroscopy

INTERVENTIONS:
Procedure: Supine Mini Percutaneous Nephrolithotomy — Percutaneous renal access and tract dilation to mini size in the supine position, followed by endoscopic stone fragmentation using laser lithotripsy, with ureteral stent placement and nephrostomy tube placement per protocol.
  Arms: Supine Mini Percutaneous Nephrolithotomy
Procedure: Flexible Ureteroscopy — Retrograde endoscopic access to the kidney using a flexible ureteroscope with laser lithotripsy for stone fragmentation, followed by ureteral stent placement per protocol.
  Arms: Flexible Ureteroscopy

SUMMARY:
This randomized controlled clinical study compared supine mini percutaneous nephrolithotomy versus flexible ureteroscopy for the management of dense lower calyceal renal stones measuring 1-2 centimeters (≤20 millimeters) with stone density greater than 1000 Hounsfield units in school-age pediatric patients aged 6-12 years. Participants were randomized to undergo either supine mini percutaneous nephrolithotomy with laser lithotripsy or flexible ureteroscopy with laser lithotripsy. The study assessed stone-free rate on non-contrast computed tomography of the urinary tract at 1 month postoperatively, along with operative time, fluoroscopy time, intraoperative and postoperative complications, and length of hospital stay. The trial has ended.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 12 years
* Single lower calyceal renal stone measuring 1-2 centimeters (≤20 millimeters) with stone density greater than 1000 Hounsfield units
* No previous urological surgery that could distort the pelvicalyceal system

Exclusion Criteria:

* Additional ureteral stones and/or congenital renal anomalies (for example, horseshoe kidney or pelviureteric junction obstruction)
* Multiple renal stones
* Untreated urinary tract infection (temporarily excluded until treated)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Stone-Free Rate | 1 month postoperatively
  Proportion of participants who were stone-free on non-contrast computed tomography of the urinary tract at 1 month after the procedure. Clinically insignificant residual fragments were defined as asymptomatic residual stones smaller than 2 millimeters.

SECONDARY OUTCOMES:
Operative Time | Intraoperative
  Total operative time for the assigned procedure (in minutes).
Fluoroscopy Time | Intraoperative
  Total fluoroscopy time used during the procedure (in seconds or minutes, per recorded operating room log).
Length of Hospital Stay | From end of procedure (day of surgery) until hospital discharge, assessed up to 30 days.
  Duration of postoperative hospital stay (in days) following the procedure.
Intraoperative and Postoperative Complications | Up to 3 months postoperatively
  Frequency and type of complications occurring intraoperatively and during follow-up after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals (Urology Department), Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data related to the primary and secondary outcomes (including demographics, baseline stone characteristics such as stone size and density, assigned intervention, operative variables, postoperative imaging results, complications, and follow-up outcomes) will be made available to qualified researchers to enable verification of results and secondary analyses. Direct identifiers will be removed, and data will be coded prior to sharing.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available beginning 6 months after study completion and will remain available for 5 years.
Access Criteria: Access will be provided upon reasonable request for research purposes. Requests must include a brief proposal and analysis plan, and investigators must agree to a data use agreement specifying: use of de-identified data only, no attempts at re-identification, no redistribution to third parties, and appropriate citation of the study. Requests should be submitted to the study team at Ain Shams University Hospitals (Urology Department) using the contact information listed in the record.